CLINICAL TRIAL: NCT01414790
Title: The Use of Human Acellular Dermal Matrix in the Prevention of Infraauricular Depressed Deformities and Frey's Syndrome Following Total Parotidectomy
Brief Title: The Use of Human Acellular Dermal Matrix to Improve Infraauricular Depressed Deformities and Frey's Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: West China Hospital of Stomatology, West China Hospital of Stomatology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: luowen228
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-01

CONDITIONS: Parotid Tumor
Keywords: human acellular dermal matrix; parotid tumor; total parotidectomy
MeSH Terms: conditions — Parotid Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADM group (Experimental): 29 patients (ADM group) had a total parotidectomy with a simultaneous ADM implantation
  Interventions: Procedure: ADM
- control group (No Intervention): 41 patients (control group) had a total parotidectomy alone

INTERVENTIONS:
Procedure: ADM — 29 patients (ADM group) had a total parotidectomy with a simultaneous ADM implantation
  Other Names: Acellular dermal matrix
  Arms: ADM group

SUMMARY:
The aim of the study was to explore whether human acellular dermal matrix (ADM) implantation could prevent infraauricular depressed deformities and Frey's syndrome following total parotidectomy.

DETAILED DESCRIPTION:
Seventy patients who underwent total parotidectomy were selected for inclusion in the study. We analyzed 41 cases of total parotidectomy (control group) and 29 cases of simultaneous ADM implantation following total parotidectomy (ADM group) for infraauricular depressed deformities and the presence of gustatory flushing or sweating. The follow-up periods ranged from 6 months to 7 years.

The Results showed facial contours and bilateral symmetry improved after surgery in the ADM group. In the control group, an infraauricular depressed deformity was evident in all 41 cases. Frey's syndrome was recorded in one patient (3.4%) from the ADM group and 14 patients (34.1%) from the control group. No cases of immune rejection, infection, hematoma, or salivary fistula were observed in either group.

ELIGIBILITY:
Inclusion Criteria:

* (1) a clinical and imaging diagnosis of either a malignant parotid tumor or deep parotid tumor
* (2) no previous surgical treatment

Exclusion Criteria:

* recurrent parotid tumors or patients who had previously undergone unsuccessful surgery

Ages: 10 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2004-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
infraauricular depressed deformities and the presence of gustatory flushing or sweating | from 6 months to 7 years after surgery
  to explore whether human acellular dermal matrix (ADM) implantation could prevent infraauricular depressed deformities and Frey's syndrome following total parotidectomy

CONTACTS AND LOCATIONS:
Overall Officials: Wen Luo, DMD, Study Chair — West China Hospital of Stomatology
Locations (1):
- West China Hospital of Stomatology, Chengdu, Sichuan, China

REFERENCES:
- [Result] Sinha UK, Saadat D, Doherty CM, Rice DH. Use of AlloDerm implant to prevent frey syndrome after parotidectomy. Arch Facial Plast Surg. 2003 Jan-Feb;5(1):109-12. doi: 10.1001/archfaci.5.1.109. PMID 12533152